CLINICAL TRIAL: NCT05872594
Title: Assessing the Prevalence and Associated Risk Factors of a Phenomenon of Epic Dream Disorder: a Cross-sectional Study
Brief Title: Prevalence of a Phenomenon of Epic Dream Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Polina Pchelina, assistant professor, I.M. Sechenov First Moscow State Medical University
Other Study IDs: 0000640001
Record Dates: First submitted 2022-09-27; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Dream Disorder
Keywords: dream; epic dream disorder; daytime symptoms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: all participants older than 18 years who agreed to participate (i.e., who clicked on the button "agree" after reading informed consent form) with no regard to sex, race, education, family status
  Interventions: Diagnostic Test: Online questionnaire

INTERVENTIONS:
Diagnostic Test: Online questionnaire — data will be collected remotely on the online platform Qualtrics

SUMMARY:
A single-center, cross-sectional, non-interventional study based on the sleep department of the Kozhevnikov Clinic for Nervous Diseases at Sechenov University. A.Y. Kozhevnikov Sechenov University is being conducted between September 2022 and December 2023 to assess the prevalence and associated symptoms and risk factors of a multiple dreams with vivid emotion, causing morning and daytime symptoms - phenomenon of Epic Dream Disorder (EDD). Demographic, sleep and psychological characteristics of people with multiple dreams will be identified, including the following standardized scales: Spielberger Anxiety Scale, Beck Depression Scale, Shortened Sleep Questionnaire. Data will be collected by mean of online questionnaire tool. According to the data obtained, prevalence of the phenomenon, differences between continuous, rank and categorical variables will be calculated in participants with and without EDD. Multivariate logistic regression will be performed to assess associated risk factors of EDD.

DETAILED DESCRIPTION:
In clinical practice, there are patients complaining for numerous dreams, which negatively affect the daytime well-being of patients, although these complaints do not fall into the category of nightmares. There are currently no data on the prevalence of the phenomenon of this phenomenon. Studies conducted on small groups of patients have found that they are more likely to have chronic pain syndrome, family history of their complaints.

The proposed study will be able to provide the first data on the prevalence and concomitant symptoms of multiple dreams. This will allow the authors to give a more precise definition of this phenomenon, describe its concomitant symptoms, and evaluate the relevance of its diagnosis and treatment. The results of the study will set the stage for further clinical research on the pathogenesis and therapy approaches. The further studies are needed to explain the causes of this phenomenon to the patients and provide them with the necessary assistance.

In view of the high workload of the medical staff, and clinical centers under the COVID-19 pandemic, and in order to increase convenience for both study participants and the researchers, data for this study will be collected remotely. The implementation of the study objectives did not require a face-to-face examination of the participants. Internet-based data collection will further simplify the processing of the data. This approach to conducting the study has already shown its applicability in a number of clinical trials.

The study will be conducted at the I.M. Sechenov First Moscow State Medical University, Russian Ministry of Health, UTH No. 3, Clinic of Nervous Diseases. A.Y. Kozhevnikov, Department of Sleep Medicine.

This study plans to inсlude all participants who agreed to participate (i.e., who clicked on the button "agree" after reading informed consent form). Information about the study and link to the questionnaires and informed consent form will be spreaded in social media, student communities, and university departmental staff communities The demographic, sleep, and psychological characteristics of people with multiple dreams will be assessed. Then a statistical analysis will be performed to compare the differences in rank, continuous, and categorical variables, and perform a multivariate logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* consent to participate in the study, expressed by ticking the appropriate box on the website after reading the text of the informed consent, confirming their understanding of the study and their consent to participate in it;

Exclusion Criteria:

* age < 18 years; This criterion is evaluated when completing the questionnaire, questionnaires from participants under 18 years old will not be included in the statistical analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Conditionally healthy individuals expressing their interest to participate by clicking the link to the questionnaires and informed consent form that will be spreaded in social media, student communities, and university departmental staff communities
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the phenomenon of epic dream disorder | Through study completion, an average of 1 year
  prevalence of the disease - the proportion of participants with the diagnosed epic dream disorder to the whole sample

SECONDARY OUTCOMES:
Demographic outcomes: Sex | Through study completion, an average of 1 year
  options (male, female)
Demographic outcomes: Age | Through study completion, an average of 1 year
  Age in years
Demographic outcomes: Weight | Through study completion, an average of 1 year
  Weight in kg
Demographic outcomes: Height | Through study completion, an average of 1 year
  Height in cm
Demographic outcomes: Level of education | Through study completion, an average of 1 year
  choose category for the level of education
Demographic outcomes: name the University | Through study completion, an average of 1 year
  For students only
Demographic outcomes: name your department | Through study completion, an average of 1 year
  For students only
Demographic outcomes: year of study | Through study completion, an average of 1 year
  For students only
Demographic outcomes: Employment status | Through study completion, an average of 1 year
  choose category for the employment status and specify your scope of activities if any
use of nicotine | Through study completion, an average of 1 year
  Fact and frequency of use of nicotine
use of alcohol | Through study completion, an average of 1 year
  Fact and frequency of use of alcohol
Medical history | Through study completion, an average of 1 year
  Presence of any chronic illnesses (specify the name)
duration of complaints | Through study completion, an average of 1 year
  Question: how long do you experience multiple dreams
Average duration of sleep | Through study completion, an average of 1 year
  hours
dreams during daytime nap | Through study completion, an average of 1 year
  Presence of dreams during daytime nap (yes or no)
Amount of dreams during the night | Through study completion, an average of 1 year
  specify number (0, 1, 2, 3 and more)
discomfort after the night of active dreaming | Through study completion, an average of 1 year
  Presence of discomfort after the night of active dreaming in the morning or during the day
triggers of active dreaming | Through study completion, an average of 1 year
  Were you able to identify a factor or event that triggered the appearance of multiple dreams? If yes, specify.
Intensity of thought activity in dream | Through study completion, an average of 1 year
  range 1-5
Intensity of speech activity in dream | Through study completion, an average of 1 year
  range 1-5
Intensity of running in dream | Through study completion, an average of 1 year
  range 1-5
Intensity of walking in dream | Through study completion, an average of 1 year
  range 1-5
Intensity of monotonous physical movements in dream | Through study completion, an average of 1 year
  range 1-5
Intensity of flight in dream | Through study completion, an average of 1 year
  range 1-5
Intensity of swimming in dream | Through study completion, an average of 1 year
  range 1-5
Intensity of jumping in dream | Through study completion, an average of 1 year
  range 1-5
Intensity of trip by transport in dream | Through study completion, an average of 1 year
  range 1-5
recalling dreams upon awakening | Through study completion, an average of 1 year
  Question: After waking up, do you remember what you saw in the dream? with 3 options - I remember that I had a dream, but I don't remember what it was about
  * I remember what the dream was about
  * I remember all the details of the dream
characteristics of dream content | Through study completion, an average of 1 year
  Intensity of positive emotions (range 1-5)
characteristics of dream content | Through study completion, an average of 1 year
  Intensity of negative emotions (range 1-5)
Impression that your brain stays awake while you sleep | Through study completion, an average of 1 year
  range 1-5
Any peculiarities of your dream | Through study completion, an average of 1 year
  specify
Awareness of a dream | Through study completion, an average of 1 year
  I don't realize I'm dreaming; I am aware that I am dreaming, but I have no control; Awareness of dreaming and controlling; I realize that I'm dreaming and I can change the plot
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptome Having difficulty knowing whether something happened in the dream or in reality
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom the feeling you had in the dream persists during the wakefulness for more than a few seconds
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Heart palpitations
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Shortness of breath
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Hyperhidrosis
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom feeling Cold
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Fatigue
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Bad mood
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Muscle pain
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Headache
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Pain in chest
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Balance disturbance
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Loss of tactile sensitivity
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Tingling/frowning sensation
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Anxiety
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Weakness
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the symptom Nausea
Subjective symptoms in the morning after a night of active dreaming | Through study completion, an average of 1 year
  Presence and length of the other symptoms, if any
Use of medications | Through study completion, an average of 1 year
  Question about the use of medication, no or yes (specify the name)
Dose of medications | Through study completion, an average of 1 year
  Question about the dose of medication, if any
Frequency of medications | Through study completion, an average of 1 year
  Question about the frequency of medications use, if any
awakenings during the night | Through study completion, an average of 1 year
  Number of awakenings during the night
Frequency of nights with multiple dreams | Through study completion, an average of 1 year
  Number of nights per week
Seasonal fluctuation of the multiple dreams | Through study completion, an average of 1 year
  During which season do the multiple dreams occur more often
Family history of Excessive dream disorder | Through study completion, an average of 1 year
  Did any of your family members has the same complaints, if yes, specify
Depression symptoms | Through study completion, an average of 1 year
  Beck Depression scale
State anxiety symptoms | Through study completion, an average of 1 year
  State anxiety by Spielberger Anxiety Scale
Trait anxiety symptoms | Through study completion, an average of 1 year
  Trait anxiety by Spielberger Anxiety Scale
Shortened Sleep Questionnaire | Through study completion, an average of 1 year
  Validated questionnaire to evaluate insomniac complaints, parasomnias, use of medications, hypersomnias, sleep related breathe disorders

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Poluektov, PhD, Study Director — I.M. Sechenov First Moscow State Medical University (Sechenov University); Polina Pchelina, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- II.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided